CLINICAL TRIAL: NCT00466271
Title: Prediction of Significant Hepatic Fibrosis in HCV Carriers With Persistently Normal Alanine Aminotransferase Levels by Splenic Arterial Pulsatility Index- A Validation Study
Brief Title: Prediction of Significant Hepatic Fibrosis in HCV Carriers With PNALT by SAPI- A Validation Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200611011R
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Chronic Hepatitis C; Hepatic Fibrosis
Keywords: Chronic hepatitis C; Persistently normal alanine aminotransferase levels; Hepatic fibrosis; Non-invasive diagnosis; Splenic arterial pulsatility index
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to validate the diagnostic accuracy and reproducibility of SAPI to predict significant hepatic fibrosis in HCV patients with PNALT who are scheduled to receive combination therapy with pegylated interferon plus ribavirin and percutaneous liver biopsies.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a major health problem, affecting 170 million persons worldwide. Approximately 25-30% of patients with chronic hepatitis C have persistently normal alanine aminotransferase (PNALT) levels, and another 40% have ALT levels less than twice the upper limit of normal (ULN). PNALT is generally defined as at least three normal ALT levels documented at least 2 months apart over a period of 6 months. Although the natural history of HCV carriers with PNALT levels remains unclear, most of them may have mild necroinflammation with mild or no fibrosis on liver histology, and the rate of disease progression is slower than patients with elevated ALT levels. However, some patients with PNALT levels still present with advanced fibrosis or even cirrhosis. A recent study has shown that combined pegylated interferon alpha plus ribavirin treatment for HCV carriers with PNALT levels can achieve comparable sustained virological response (SVR) to those with elevated ALT levels, suggesting antiviral therapy could be initiated irrespective of ALT levels. Furthermore, patients with initial diagnosis of significant fibrosis on liver biopsies harbor higher risks to advanced fibrosis and cirrhosis, and may merit antiviral therapy to stop or delay the progression of hepatic fibrosis.

Currently, liver biopsy is recognized as the gold standard for assessing the grade of necroinflammation and stage of fibrosis before the initiation of antiviral therapy. However, it is costly and harbors risk of complications. In addition, sampling error due to the non-uniform distribution of the parenchymal damage, as well as intra- and inter-observer variability is often encountered. A noninvasive tool to evaluate liver disease activity or fibrosis stage is helpful, particularly in monitoring HCV carriers over time.

Studies assessing the usefulness of noninvasive tests to predict hepatic fibrosis were mainly performed in patients with elevated ALT levels. In patients with PNALT levels, only three studies have addressed the value of Fibroscan, Fibro Test and aspartate aminotransferase (AST) to platelet ratio index (APRI). However, Fibro Test is costly and Fibroscan has not been widely used. In addition, APRI has not been shown by other cohorts in patients with PNALT levels to possess excellent diagnostic accuracy and reproducibility (32). Currently, splenic arterial pulsatility index (SAPI) has been shown to have superior diagnostic accuracy to various biochemical indices (including APRI, API (age-platelet index), and AAR (AST to ALT ratio)) in predicting significant hepatic fibrosis in HCV carriers with PNALT. However, SAPI has not been validated in an independently prospective cohort to confirm both the diagnostic accuracy and reproducibility. Therefore, our study is aimed to validate the diagnostic accuracy and reproducibility of SAPI to predict significant hepatic fibrosis in HCV patients with PNALT who are scheduled to receive combination therapy with pegylated interferon plus ribavirin and percutaneous liver biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* HCV RNA and anti-HCV positivity for more than 6 months
* 4 consecutive normal ALT values (< 40 IU/L for men and < 34 IU/L for women)at 3 months apart over a period of 12 months

Exclusion Criteria:

* HBV and HCV co-infection
* HBV and HIV co-infection
* History of heavy alcohol use (> 50 gram/day)
* Autoimmune liver diseases
* Metabolic liver diseases
* Presence of hepatocellular carcinoma
* Bleeding tendency
* Decline liver biopsies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV carriers with persistently normal ALT levels who will receive percutaneous liver biopsy
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Director — Department of Internal Medicine, National Taiwan Universitys Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Bacon BR. Treatment of patients with hepatitis C and normal serum aminotransferase levels. Hepatology. 2002 Nov;36(5 Suppl 1):S179-84. doi: 10.1053/jhep.2002.36386. PMID 12407592
- [Background] EASL International Consensus Conference on Hepatitis C. Paris, 26-28, February 1999, Consensus Statement. European Association for the Study of the Liver. J Hepatol. 1999 May;30(5):956-61. No abstract available. PMID 10365827
- [Background] Puoti C, Guido M, Mangia A, Persico M, Prati D; Committee on HCV carriers with normal alanine aminotransferase levels of the Italian Association for the Study of the Liver. Clinical management of HCV carriers with normal aminotransferase levels. Dig Liver Dis. 2003 May;35(5):362-9. doi: 10.1016/s1590-8658(03)00185-3. PMID 12846410
- [Background] Gholson CF, Morgan K, Catinis G, Favrot D, Taylor B, Gonzalez E, Balart L. Chronic hepatitis C with normal aminotransferase levels: a clinical histologic study. Am J Gastroenterol. 1997 Oct;92(10):1788-92. PMID 9382037
- [Background] Puoti C, Magrini A, Stati T, Rigato P, Montagnese F, Rossi P, Aldegheri L, Resta S. Clinical, histological, and virological features of hepatitis C virus carriers with persistently normal or abnormal alanine transaminase levels. Hepatology. 1997 Dec;26(6):1393-8. doi: 10.1053/jhep.1997.v26.pm0009397976.
- [Background] Conry-Cantilena C, VanRaden M, Gibble J, Melpolder J, Shakil AO, Viladomiu L, Cheung L, DiBisceglie A, Hoofnagle J, Shih JW, et al. Routes of infection, viremia, and liver disease in blood donors found to have hepatitis C virus infection. N Engl J Med. 1996 Jun 27;334(26):1691-6. doi: 10.1056/NEJM199606273342602. PMID 8637513
- [Background] Pradat P, Alberti A, Poynard T, Esteban JI, Weiland O, Marcellin P, Badalamenti S, Trepo C. Predictive value of ALT levels for histologic findings in chronic hepatitis C: a European collaborative study. Hepatology. 2002 Oct;36(4 Pt 1):973-7. doi: 10.1053/jhep.2002.35530. PMID 12297846
- [Background] Alberti A, Noventa F, Benvegnu L, Boccato S, Gatta A. Prevalence of liver disease in a population of asymptomatic persons with hepatitis C virus infection. Ann Intern Med. 2002 Dec 17;137(12):961-4. doi: 10.7326/0003-4819-137-12-200212170-00009. PMID 12484711
- [Background] Persico M, Persico E, Suozzo R, Conte S, De Seta M, Coppola L, Palmentieri B, Sasso FC, Torella R. Natural history of hepatitis C virus carriers with persistently normal aminotransferase levels. Gastroenterology. 2000 Apr;118(4):760-4. doi: 10.1016/s0016-5085(00)70145-4. PMID 10734027
- [Background] Martinot-Peignoux M, Boyer N, Cazals-Hatem D, Pham BN, Gervais A, Le Breton V, Levy S, Degott C, Valla DC, Marcellin P. Prospective study on anti-hepatitis C virus-positive patients with persistently normal serum alanine transaminase with or without detectable serum hepatitis C virus RNA. Hepatology. 2001 Nov;34(5):1000-5. doi: 10.1053/jhep.2001.28458. PMID 11679971
- [Background] Mathurin P, Moussalli J, Cadranel JF, Thibault V, Charlotte F, Dumouchel P, Cazier A, Huraux JM, Devergie B, Vidaud M, Opolon P, Poynard T. Slow progression rate of fibrosis in hepatitis C virus patients with persistently normal alanine transaminase activity. Hepatology. 1998 Mar;27(3):868-72. doi: 10.1002/hep.510270333. PMID 9500720
- [Background] Jamal MM, Soni A, Quinn PG, Wheeler DE, Arora S, Johnston DE. Clinical features of hepatitis C-infected patients with persistently normal alanine transaminase levels in the Southwestern United States. Hepatology. 1999 Nov;30(5):1307-11. doi: 10.1002/hep.510300526. PMID 10534355
- [Background] Okanoue T, Makiyama A, Nakayama M, Sumida Y, Mitsuyoshi H, Nakajima T, Yasui K, Minami M, Itoh Y. A follow-up study to determine the value of liver biopsy and need for antiviral therapy for hepatitis C virus carriers with persistently normal serum aminotransferase. J Hepatol. 2005 Oct;43(4):599-605. doi: 10.1016/j.jhep.2005.04.008. PMID 16024129
- [Background] Hui CK, Belaye T, Montegrande K, Wright TL. A comparison in the progression of liver fibrosis in chronic hepatitis C between persistently normal and elevated transaminase. J Hepatol. 2003 Apr;38(4):511-7. doi: 10.1016/s0168-8278(03)00004-7. PMID 12663245
- [Background] Zeuzem S, Diago M, Gane E, Reddy KR, Pockros P, Prati D, Shiffman M, Farci P, Gitlin N, O'Brien CB, Lamour F, Lardelli P; PEGASYS Study NR16071 Investigator Group. Peginterferon alfa-2a (40 kilodaltons) and ribavirin in patients with chronic hepatitis C and normal aminotransferase levels. Gastroenterology. 2004 Dec;127(6):1724-32. doi: 10.1053/j.gastro.2004.09.050. PMID 15578510
- [Background] Piccinino F, Sagnelli E, Pasquale G, Giusti G. Complications following percutaneous liver biopsy. A multicentre retrospective study on 68,276 biopsies. J Hepatol. 1986;2(2):165-73. doi: 10.1016/s0168-8278(86)80075-7. PMID 3958472
- [Background] Cadranel JF, Rufat P, Degos F. Practices of liver biopsy in France: results of a prospective nationwide survey. For the Group of Epidemiology of the French Association for the Study of the Liver (AFEF). Hepatology. 2000 Sep;32(3):477-81. doi: 10.1053/jhep.2000.16602. PMID 10960438
- [Background] McGill DB, Rakela J, Zinsmeister AR, Ott BJ. A 21-year experience with major hemorrhage after percutaneous liver biopsy. Gastroenterology. 1990 Nov;99(5):1396-400. doi: 10.1016/0016-5085(90)91167-5. PMID 2101588
- [Background] Maharaj B, Maharaj RJ, Leary WP, Cooppan RM, Naran AD, Pirie D, Pudifin DJ. Sampling variability and its influence on the diagnostic yield of percutaneous needle biopsy of the liver. Lancet. 1986 Mar 8;1(8480):523-5. doi: 10.1016/s0140-6736(86)90883-4. PMID 2869260
- [Background] Bedossa P, Dargere D, Paradis V. Sampling variability of liver fibrosis in chronic hepatitis C. Hepatology. 2003 Dec;38(6):1449-57. doi: 10.1016/j.hep.2003.09.022. PMID 14647056
- [Background] Colloredo G, Guido M, Sonzogni A, Leandro G. Impact of liver biopsy size on histological evaluation of chronic viral hepatitis: the smaller the sample, the milder the disease. J Hepatol. 2003 Aug;39(2):239-44. doi: 10.1016/s0168-8278(03)00191-0. PMID 12873821
- [Background] Giannini E, Risso D, Botta F, Chiarbonello B, Fasoli A, Malfatti F, Romagnoli P, Testa E, Ceppa P, Testa R. Validity and clinical utility of the aspartate aminotransferase-alanine aminotransferase ratio in assessing disease severity and prognosis in patients with hepatitis C virus-related chronic liver disease. Arch Intern Med. 2003 Jan 27;163(2):218-24. doi: 10.1001/archinte.163.2.218. PMID 12546613
- [Background] Imbert-Bismut F, Ratziu V, Pieroni L, Charlotte F, Benhamou Y, Poynard T; MULTIVIRC Group. Biochemical markers of liver fibrosis in patients with hepatitis C virus infection: a prospective study. Lancet. 2001 Apr 7;357(9262):1069-75. doi: 10.1016/S0140-6736(00)04258-6. PMID 11297957
- [Background] Poynard T, Bedossa P. Age and platelet count: a simple index for predicting the presence of histological lesions in patients with antibodies to hepatitis C virus. METAVIR and CLINIVIR Cooperative Study Groups. J Viral Hepat. 1997 May;4(3):199-208. doi: 10.1046/j.1365-2893.1997.00141.x. PMID 9181529
- [Background] Wai CT, Greenson JK, Fontana RJ, Kalbfleisch JD, Marrero JA, Conjeevaram HS, Lok AS. A simple noninvasive index can predict both significant fibrosis and cirrhosis in patients with chronic hepatitis C. Hepatology. 2003 Aug;38(2):518-26. doi: 10.1053/jhep.2003.50346. PMID 12883497
- [Background] Castera L, Vergniol J, Foucher J, Le Bail B, Chanteloup E, Haaser M, Darriet M, Couzigou P, De Ledinghen V. Prospective comparison of transient elastography, Fibrotest, APRI, and liver biopsy for the assessment of fibrosis in chronic hepatitis C. Gastroenterology. 2005 Feb;128(2):343-50. doi: 10.1053/j.gastro.2004.11.018. PMID 15685546
- [Background] Colletta C, Smirne C, Fabris C, Toniutto P, Rapetti R, Minisini R, Pirisi M. Value of two noninvasive methods to detect progression of fibrosis among HCV carriers with normal aminotransferases. Hepatology. 2005 Oct;42(4):838-45. doi: 10.1002/hep.20814. PMID 16121354
- [Background] Sebastiani G, Vario A, Guido M, Noventa F, Plebani M, Pistis R, Ferrari A, Alberti A. Stepwise combination algorithms of non-invasive markers to diagnose significant fibrosis in chronic hepatitis C. J Hepatol. 2006 Apr;44(4):686-93. doi: 10.1016/j.jhep.2006.01.007. Epub 2006 Feb 8. PMID 16490278
- [Background] Fabris C, Smirne C, Toniutto P, Colletta C, Rapetti R, Minisini R, Falleti E, Pirisi M. Assessment of liver fibrosis progression in patients with chronic hepatitis C and normal alanine aminotransferase values: the role of AST to the platelet ratio index. Clin Biochem. 2006 Apr;39(4):339-43. doi: 10.1016/j.clinbiochem.2006.01.011. Epub 2006 Feb 20. PMID 16487951
- [Result] Liu CH, Lin JW, Tsai FC, Yang PM, Lai MY, Chen JH, Kao JH, Chen DS. Noninvasive tests for the prediction of significant hepatic fibrosis in hepatitis C virus carriers with persistently normal alanine aminotransferases. Liver Int. 2006 Nov;26(9):1087-94. doi: 10.1111/j.1478-3231.2006.01355.x. PMID 17032409